CLINICAL TRIAL: NCT06143462
Title: The Effect of Vestibular Rehabilitation Treatment (VRT) on Patients With Unsteadiness After Intratympanic Gentamicin in Meniere's Disease: Protocol for a Randomized Controlled Trial
Brief Title: Vestibular Rehabilitation for Unsteadiness After Intratympanic Gentamicin in Patients With Meniere's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202311-MD-ITG-VRT
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: usual care (UC) (Active Comparator): Group A (UC) will receive conventional medications.
  Interventions: Drug: Usual care; Other: Health Education
- Group B: vestibular rehabilitation treatment (VRT) (Experimental): Group B (VRT) will receive outpatient VRT in combination with home practice based on conventional treatment.
  Interventions: Behavioral: vestibular rehabilitation

INTERVENTIONS:
Drug: Usual care — Include anti-dizziness medications, diuretics, or hormone therapy.
  Arms: Group A: usual care (UC)
Other: Health Education — Include comprehensive health education, fall prevention and lifestyle adjustments.
  Arms: Group A: usual care (UC)
Behavioral: vestibular rehabilitation — Encompass office-based sessions of vestibular rehabilitation treatment once weekly, supplemented by home-based exercises conducted two or three times daily for the remaining duration of the study.
  Arms: Group B: vestibular rehabilitation treatment (VRT)

SUMMARY:
To investigate the efficacy of vestibular rehabilitation treatment on unsteadiness after intratympanic gentamicin in patients with Meniere's disease.

DETAILED DESCRIPTION:
Previous studies have generally focused on the efficacy of VRT for Meniere's disease, with little attention paid to the effect of VRT on MD patients who still have vestibular dysfunction even after intratympanic gentamicin treatment.

The aim of this study is to compare the efficacy of VRT with usual care in MD patients who experience persistence of unsteadiness 1 month after intratympanic gentamicin treatment, in order to understand whether VR has a positive impact on balance maintenance and vertigo control in MD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 75 years old;
2. Complained of persistent unsteadiness 1 month after intratympanic gentamicin treatment;
3. Be willing to sign the informed consent of the study.

Exclusion Criteria:

1. Conformed to neuromuscular disease;
2. Conformed to severe cervical spine disease;
3. Conformed to congenital inner ear disease (except vestibular migraine(VM))
4. Concurrent manifestation of psychiatric or psychological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Gait Assessment (FGA) | Change from baseline, at 8 weeks and 6 months post-randomization
  FGA is a semi-quantitative measure of walking balance ability.

SECONDARY OUTCOMES:
Sensory Organization Test (SOT) | Change from baseline, at 8 weeks and 6 months post-randomization
  SOT is a form of posturography, aiming to distinguish and assess the weight of vestibular, visual, and proprioceptive sensations in maintaining balance.
Meniere's Disease Outcomes Questionnaire (MDOQ) | Change from baseline, at 8 weeks and 6 months post-randomization
  MDOQ is a comprehensive assessment of MD patients' quality of life (QOL) in three dimensions: physical, emotional, and social.
Visual Vertigo Analogue Scale (VVAS) | Change from baseline, at 8 weeks and 6 months post-randomization
  In VVAS, patients estimate the intensity of their symptoms related to dizziness, vertigo, and imbalance.
Vestibular Activities and Participation Measure (VAP) | Change from baseline, at 8 weeks and 6 months post-randomization
  VAP is a 34-item self-report questionnaire, aiming to evaluate the extent of activity limitations and participation restrictions created by vestibular disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqian Yu, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Tong Q, Zhou Y, Wu P, Yu H. Effect of vestibular rehabilitation treatment (VRT) on patients with unsteadiness after intratympanic gentamicin in Meniere's disease: protocol for a randomised controlled trial. BMJ Open. 2025 Feb 22;15(2):e088722. doi: 10.1136/bmjopen-2024-088722. PMID 39987011